CLINICAL TRIAL: NCT06831006
Title: A Randomized Controlled Trial (RCT) Evaluating the Effects of Cool Roofs on Health Outcomes Using Smartwatches in Hermosillo, Mexico
Brief Title: Assessing the Effect of Cool Roofs on Health Using Smartwatches in Hermosillo, Mexico
Acronym: REFLECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Heidelberg University (Other); London School of Hygiene and Tropical Medicine (Other); Rutgers University (Other); Instituto Tecnológico de Hermosillo (Unknown); Labfront (Industry); Wellcome Trust (Other); Hermosillo City Government (Unknown); EPS (Unknown)
Responsible Party: Principal Investigator, Aditi Bunker, Principal Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728165; 226745/Z/22/Z (Other Grant/Funding Number: Wellcome Trust UK)
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Heart Rate; All-day Steps; Distance Walked; Active Minutes; Moderate-intensity Activity Minutes; Vigorous-intensity Activity Duration; Sleep Quantity; Time in Sleep Stages; Awake Duration; Sleep Score
Keywords: Hot Temperature; Humidity; Housing; Wearable; Smartwatch; Heart rate; Cardiovascular; Physical activity; Sleep; Cool roof; Heat stress
MeSH Terms: conditions — Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cool roof (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- No cool roof (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a heat-reflecting material that can be applied to existing household roofing in the form of a liquid-applied membrane. Cool roofs work by increasing solar reflectance (the ability to reflect the visible wavelengths of sunlight, reducing heat transfer to the surface) and thermal emittance (the ability to radiate absorbed solar energy) thereby reducing the amount of heat transferred into the home.
  Arms: Cool roof

SUMMARY:
Ambient air temperatures in Mexico have broken record highs in 2024 with Hermosillo reaching the highest maximum temperature recorded in Mexico at 51.9 C. Solutions are needed to build heat resilience in communities and adapt to increasing heat from climate change. Sunlight-reflecting cool roof coatings may passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions in the northern zone of Mexico are susceptible to increased heat exposure.

Heat exposure can instigate and worsen numerous physical, mental and social health conditions. The worst adverse health effects are experienced in communities that are least able to adapt to heat exposure. By reducing indoor temperatures, cool roof use may promote heart health, sleep and physical activity in household occupants.

The long-term research goal of the investigators is to identify viable passive housing adaptation technologies with proven health benefits to reduce the burden of heat stress in communities affected by heat in northern zone of Mexico. To meet this goal, the investigators will conduct a randomized controlled trial to establish the effects of cool roof use on heart rate, sleep and physical activity in Hermosillo, Mexico.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low-resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen health conditions, including cardiovascular, metabolic, endocrine and respiratory disease, heat-related illnesses, pregnancy complications, and mental health conditions. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially homes, is ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, there currently is a lack of evidence on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce heat stress in low-resource settings.

Cities and towns of LMIC are among the most vulnerable to the adverse impacts of climate change and are likely to experience increases in ambient air temperature over the coming decades. People in Hermosillo (located in the State of Sonora, Mexico) are exposed to heat and low humidity year-round. The State of Sonora has a large burden of non-communicable diseases (NCDs), with nearly 28% of deaths due to NCDs, such as heart diseases and diabetes mellitus. The combined burden of heat and NCDs places Sonora's, especially Hermosillo's, populations at greater risk of adverse health effects from heat extremes.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. The investigators therefore aim to conduct a randomized controlled trial investigating the effects of cool roofs on heart rate, sleep and physical activity using smartwatches in Hermosillo.

The trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in Hermosillo. Findings will inform regional and global policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

* Permanent household resident

Exclusion Criteria:

* Roof damage, inaccessible or instability of roof adversely affecting cool roof coating application.
* Participant unable to provide written/verbal informed consent. Participants will be excluded if they are not willing or able to wear a smartwatch.
* Participants will be excluded if they do not have a smartphone with an internet connection that can connect to the smartwatch.
* Only one participant per household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Heart rate in beats per minute measured at 15-second intervals using Garmin Vivosmart 5 devices.

SECONDARY OUTCOMES:
All-day steps | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of steps measured daily using Garmin Vivosmart 5 devices.
Active minutes | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of active exercise daily using Garmin Vivosmart 5 devices.
Distance walked | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total distance walked daily using Garmin Vivosmart 5 devices.
Moderate-intensity activity minutes | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at barements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of moderate-intensity activity daily using Garmin Vivosmart 5 devices.
Vigorous-intensity activity duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of vigorous-intensity activity daily using Garmin Vivosmart 5 devices.
Sleep quantity | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent asleep each night using Garmin Vivosmart 5 devices.
Time in sleep stages | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent in sleep stages each night using Garmin Vivosmart 5 devices.
Awake duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent awake during sleep time each night using Garmin Vivosmart 5 devices.
Sleep score | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The Garmin sleep score (0-100) each night using Garmin Vivosmart 5 devices. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Tukuitonga, Sir. Dr., Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Instituto Tecnológico de Hermosillo, Hermosillo, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers. Individual names of study participants and identifying factors will be removed prior to data sharing.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication.
URL: http://reflect.org.nz